CLINICAL TRIAL: NCT03927729
Title: Use of Methoxyflurane (Penthrox) as an Antalgic in Hospital Trauma
Acronym: UMATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DR190096; 2019-A00259-48 (Other: IdRCB)
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Pain; Traumatic Injury
Keywords: Methoxyflurane; Penthrox; non opioid analgesia; traumatic pain; pain; antalgic protocol; emergency department
MeSH Terms: conditions — Pain; Wounds and Injuries; Emergencies | interventions — Methoxyflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penthrox (Experimental): Patients with moderate to severe post-traumatic acute pain will be included in the emergency room.
  Interventions: Drug: Methoxyflurane

INTERVENTIONS:
Drug: Methoxyflurane — Pain will be treated with inhaled methoxyflurane (Penthrox®).
  Other Names: Penthrox®)

SUMMARY:
Study of traumatized patients treated in emergency departments of Tours, seeking to optimize the management of trauma pain in an inpatient setting, with the opportunity to integrate inhaled methoxyflurane (Penthrox®) into the arsenal analgesics useful in the analgesic protocol of the Reception and Orientation Nurse.

DETAILED DESCRIPTION:
Intra-hospital, the prevalence of pain is major; this is variable depending on the studies, but permanently above 60%. A study conducted in 2015 in Tours Adult Emergencies showed a prevalence of pain of 66.5% with an average waiting time of 2h28 before receiving an analgesic.

The pain management protocol at the Tours emergency department includes paracetamol for a numerical evaluation scale (EN) < 3 and tramadol for an EN between 4 and 6. But these therapies have a delay of action too long or are given too late. An improvement in the management of pain in emergency is therefore necessary.

Methoxyflurane (Penthrox®) is a volatile fluoridated analgesic; it offers several benefits: fast over a long period, well tolerated, effective and without interference with other drugs. Despite a misuse in the 70s, it has been used for more than 20 years in Australia and New Zealand. It was granted marketing authorization in 2016 and has been marketed in France since 2017.

It should be noted that this analgesic treatment is already adopted in several hospitals in the region and also in the SAMU 37.

A similar study was conducted in Grenoble but on a different population. The investigators plan to highlight the interest of Penthrox® in the management of monotraumatic pains in the Adult Emergencies of Tours with the intention of modifying the antalgic protocol accordingly to the reception of emergencies.

ELIGIBILITY:
Inclusion Criteria:

* Conscious patient
* Age ≥ 18 years
* Acute pain of monotraumatic origin
* Pain > 4 on a visual numerical scale

Exclusion Criteria:

* State of shock with unstable hemodynamics (PA <90/60)
* Suspected or proven trauma to the chest, abdomen or pelvis
* Serious head trauma
* Consciousness disorder with Glasgow score <15
* Patient who has already received analgesics (with the exception of paracetamol)
* Patient receiving an intravenous approach for analgesia
* Renal or hepatic disorders known
* Hypersensitivity to fluoridated anesthetics or history of malignant hyperthermia in the patient or family
* Pregnant or nursing woman
* Patient under judicial protection
* Non communicating patient or with difficulties of understanding

Exclusion Criteria:

* Intravenous injection for analgesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
Change of traumatic acute pain level between baseline and 15 minutes | baseline and 15 minutes
  Efficiency will be measured by its effect on pain according to a visual numerical scale (VNS: between 0 and 10)

SECONDARY OUTCOMES:
Change of traumatic acute pain level between baseline and 30 minutes | baseline and 30 minutes
  Efficiency will be measured by its effect on pain according to a visual numerical scale (VNS: between 0 and 10).
Change of traumatic acute pain level between baseline and 45 minutes | baseline and 45 minutes
  Efficiency will be measured by its effect on pain according to a visual numerical scale (VNS: between 0 and 10).
Change of traumatic acute pain level between baseline and 60 minutes | baseline and 60 minutes
  Efficiency will be measured by its effect on pain according to a visual numerical scale (VNS: between 0 and 10).
Pain extinction duration | baseline and 15, 30, 45, 60 minutes
  Duration before pain extinction, evaluated using a visual numerical scale (VNS: between 0 and 10)
Penthrox tolerance | 60 minutes
  Collection of side effects
Medical team level of satisfaction | 60 minutes
  5 grades satisfaction scale filled by the medical team 30 minutes after the treatment (Very satisfied, Satisfied, Neutral, Dissatisfied, Very dissatisfied)
Patient level of satisfaction | 60 minutes
  5 grades satisfaction scale filled by the patient 30 minutes after the treatment (Very satisfied, Satisfied, Neutral, Dissatisfied, Very dissatisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Julien CONRAS, MD, Principal Investigator — University Hospital, Tours
Locations (1):
- Emergency Medical Service, University Hospital, Tours, Tours, France